CLINICAL TRIAL: NCT02091258
Title: Tooth Loss in Periodontitis Patients on Long-term Maintenance in Private Practice
Brief Title: Tooth Loss in Periodontitis Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: UCL 14/0110
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2015-09

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Tooth loss in periodontitis patients is associated with patient and site factors as well as with treatment provided. Not much is known about long-term tooth loss in periodontitis patients in private practice in the UK. The study plans to follow-up 200 subjects with periodontitis (and currently on maintenance therapy) for 5 years. The effect of treatment provided, site and patient risk factors on tooth loss will be studied.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Initial diagnosis of chronic or aggressive periodontitis (Lindhe et al. 1999, Lang et al. 1999), with at least two sites with PPD and CAL ≥5mm
2. Diagnosed and treated by the same periodontist (LN)
3. Willing to give written informed consent for study participation
4. Willing to undergo SPT as per standard of care for at least 5 years

EXCLUSION CRITERIA:

1. Serious medical history that prevents patients from undergoing dental treatment
2. History of rheumatic fever, heart murmur, mitral valve prolapse, artificial heart valve or other conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures
3. Current alcohol or drug abuse
4. Self-reported pregnancy or lactation
5. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may compromise trial participation and/or interpretation of trial results and, in the judgement of the investigator, would make the subject inappropriate for entry into this trial

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 200 patients with periodontitis on maintenance therapy (after initial/ corrective periodontal therapy) will be included in the study
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-06; Primary Completion 2020-05 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Tooth loss | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Nibali, PhD, Principal Investigator — UCL
Locations (2):
- United Kingdom (2):
  - The Dentist, Bishop's Stortford, Herts
  - Ravenscourt Dental Practice, London